CLINICAL TRIAL: NCT03531684
Title: Clinical Trial to Test the Efficacy and Safety of MMFS-205 in Early Alzheimer's Disease Patients
Brief Title: Efficacy and Safety of MMFS in Early AD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurocentria, Inc. (Industry)
Collaborators: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: NC007
Record Dates: First submitted 2018-04-04; First posted 2018-05-22 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — threonic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MMFS-205-SR (Experimental): Oral MMFS-205-SR twice daily (2,000, 3,000, or 4,000 mg/day total, depending on lean body mass and response to initial dose at Week 12) for 24 weeks
  Interventions: Dietary Supplement: MMFS-205-SR
- Placebo (Placebo Comparator): Oral inactive placebo twice daily for 24 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: MMFS-205-SR — Twice daily, oral, 500 mg tablets
  Other Names: L-threonic acid magnesium salt, L-TAMS
  Arms: MMFS-205-SR
Dietary Supplement: Placebo — Twice daily, oral
  Other Names: Inactive sugar pill
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the safety and efficacy of MMFS for improving cognition and global function in patients with probable Early Alzheimer's disease.

DETAILED DESCRIPTION:
This is a phase 2 study in patients with probable Early Alzheimer's disease (AD). Early AD includes Stage 3 AD patients (MCI due to AD) and Stage 4 AD patients (mild AD). The study is a randomized, double-blind, placebo controlled, parallel group design, in which participants (up to 6 per arm; 12 total) will receive oral placebo or MMFS twice daily for 24 weeks. Randomized patients and their informants (required) will complete 3 assessments total: at baseline (prior to taking any study tablets), week 12, and week 24 visits. At each of the three visits, participants will complete cognitive and behavioral measures and clinical interviews, a blood sample will be collected for safety and biomarkers related to Alzheimer's disease, and the informant will complete an interview concerning the patient's cognition, mood, and function. A range of safety and tolerability assessments will also be performed (including vital signs, laboratory tests, and ECGs). Participants will be contacted by phone between clinical assessments for monitoring.

ELIGIBILITY:
Inclusion Criteria

Patients meeting all of the following inclusion criteria should be considered for admission to the study:

1. MMSE ≥ 19
2. ≥ 55 and ≤ 85 years old at Screening
3. Meet criteria for at least one of the following Stages of Early Alzheimer's Disease as defined below:

   Stage 3 AD (MCI due to AD)
   1. CDR Global score = 0.5, with

      * 0.5 on memory box score; and
      * 0.5 on at least one of the following functional measures: community affairs, home & hobbies, or personal care
   2. MMSE ≥ 24

   Stage 4 AD (Mild AD):
   1. CDR Global score = 1, with

      * 0.5 on memory box score; and
      * 0.5 on at least one of the following functional measures: community affairs, home & hobbies, or personal care; OR
   2. CDR Global score = 0.5, with

      * 0.5 on memory box score; and
      * 0.5 on at least one of the following functional measures: community affairs, home & hobbies, or personal care; and MMSE 19-23
4. ≥ 3 on at least one of the following Neuropsychiatric Inventory (NPI) behavioral areas: Agitation/Aggression, Depression/Dysphoria, Anxiety, Apathy/Indifference, Disinhibition, or Irritability/Lability, and total NPI score in these behavioral areas ≥ 6.
5. Total Body weight (bw) must be ≥50 kg and ≤110 kg and lean body mass (LBM) must be ≤ 85 kg at screening
6. Must be fluent in English
7. Must have a friend/family member who frequently spends time with the subject (≥10 hours per week), and is willing to serve as an informant, and accompany the subject to, and participate in, all clinic visits
8. Completion of at least 10 years of formal education (i.e., possess high school diploma, GED, or equivalent)
9. Hearing and Vision ability sufficient to complete neurocognitive testing
10. Be able and willing to collect urine (at home) for 12 hours the day prior to follow up visits (optional for Stage 4 patients).

Exclusion Criteria

Patients meeting any of the following exclusion criteria will not be enrolled in the study:

Exclusions to rule out subjects with cognitive impairment likely due to something other than AD:

1. Known negative biomarker for brain amyloid pathology as indicated by either amyloid PET or CSF assessment or both
2. Stroke or Transient Ischemic Attack (TIA) or unexplained loss of consciousness in the past 1 year
3. Clinically significant psychiatric illness in past 6 months requiring hospitalization
4. Seizure in the past 3 years
5. Within 1 year before the screening or between screening and baseline, any of the following: myocardial infarction; moderate or severe congestive heart failure, New York Heart Association class III or IV; hospitalization for, or symptom of, unstable angina; syncope due to orthostatic hypotension or unexplained syncope; known significant structural heart disease (e.g., significant valvular disease, hypertrophic cardiomyopathy), or hospitalization for arrhythmia; congenital QT prolongation
6. Subject report of human immunodeficiency virus (HIV) infection
7. History of evidence of acute or sub-acute micro or macrohemorrhage, greater than 4 microhemorrhages, cortical infarct, or greater than one 1 lunar infarct
8. Alcohol or substance abuse in past 1 year
9. Untreated and/or uncontrolled hypothyroidism
10. Evidence of vascular dementia (Modified Hachinski Ischemia Scale score >5)
11. History of clinically important carotid or vertebrobasilar stenosis or plaque
12. Systemic chemotherapy in past 1 year
13. Diagnosis of Multiple Sclerosis
14. Unintentional rapid weight loss (>10% body weight within past 12 months)

    Exclusions to rule out subjects with potential issues absorbing or metabolizing MMFS:
15. Poor kidney function; corrected estimated glomerular filtration rate (eGFRcorr) < 40 mL/min/m2
16. History of significant gastrointestinal disorder, such as chronic Diarrhea, irritable bowel syndrome, ulcerative colitis, Chron's disease, etc.

    Exclusions to rule out subjects with sleeping problems not related to CNS disorder:
17. Diagnosed with apnea/hypopnea but not using Continuous Positive Airway Pressure (CPAP) or Bilevel Positive Airway Pressure (BIPAP). If diagnosed with apnea/hypopnea, subject must maintain use of device throughout study
18. Untreated nocturia that affects sleep

    Exclusions to rule out subjects with conditions that could affect their safety:
19. Females of child-bearing potential, as defined as menstruation within past 12 months or not surgically sterile.
20. Systolic blood pressure > 150 mm Hg
21. An affirmative response on the C-SSRS, indicating suicidal ideation with intent, with or without a plan or method, or suicidal behavior, in the past 6 months.

    Exclusions to rule out subjects with conditions that could inhibit or confound the effects of MMFS or the ability of the subject to complete the study:
22. Serious or unstable clinically important systemic illness or disease that, in the judgment of the investigator, is likely to affect cognitive assessment, deteriorate, or affect the participant's safety or ability to complete the study, including hepatic, renal, gastroenterologic, respiratory, cardiovascular, endocrinologic, immunologic, or hematologic disorders
23. Currently living in an institutional facility such as a nursing home
24. History or diagnosis of any of the following sleep conditions:

    1. Narcolepsy
    2. Cataplexy (familial or idiopathic)
    3. Circadian Rhythm Sleep Disorder
    4. Primary Hypersomnia
25. Severe physical disability not associated with cognitive function that limits ability to complete neurocognitive testing (e.g., severe tremor, debilitating arthritis)
26. Changes in medications or doses of medication in past 30 days prior to Screening

    1. All allowed concomitant medications, supplements, or other substances (with the exception of sleep, mood, cognitive and neuropsychiatric drugs) must be at stable doses for at least 30 days prior to screening and must be kept as stable as medically possible during the trial. Dosing change of ConMeds within 30 days of Screening may be allowed if in the opinion of the investigator, will not affect or influence study results.
    2. If a change in medication dosage occurs during the study, this will lead to discontinuation from study participation unless it relates to a medication that, in the view of the study investigator, does not affect participation in the trial.
    3. Allowed Sleep, Neuropsychiatric and Cognitive drugs must be stable for 90 days prior to Screening. Dosing change of Neuropsychiatric and Cognitive drugs within 90 days of Screening may be allowed if in the opinion of the investigator, will not affect or influence study results.
27. Use of prohibited medications/substances.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2020-04-22 (Actual); Study Completion 2020-04-22 (Actual)

PRIMARY OUTCOMES:
Neuropsychological Test Battery (NTB) standardized composite score | Change from baseline at 24 weeks
  Standardized composite score generated from a battery of 4 cognitive tests, including: 1) COWAT - Category Fluency assessment of semantic fluency; 2) WAIS-IV Coding (Digit Symbol Substitution Test; DSST) assesment of attention speed of processing, mental flexibility and executive function; 3) Free and Cued Selective Reminding Test Immediate Recall (FCSRT-IR) assessment of episodic visual memory; 4) Wechsler Logical Memory II (Delayed Recall) assessment of narrative memory.
Clinical Dementia Rating Scale - Sum of Boxes (CDR-SB) score | Change from baseline at 24 weeks
  Composite measure of cognition and global function. The scores in each domain range from 0-3, referring to impairment with 0 being none, 0.5 being questionable, 1 being mild, 2 being moderate, and 3 being severe.

SECONDARY OUTCOMES:
Modified Mini-Mental State Examination (mMMSE) total score | Change from baseline at 12 and 24 weeks
  Cognitive test; the mMMSE is scored as the number of correctly completed items, with lower scores indicative of poorer performance and greater cognitive impairment. The score ranges from 0 to 100, with 100 being perfect performance. An mMMSE-derived MMSE score ranging from 0 to 30, with 30 being perfect performance, can also be generated.
Alzheimer's Disease Cooperative Scale-Activities of Daily Living-Mild Cognitive Impairment 24 questions (ADCS-ADL-MCI24) | Change from baseline at 12 and 24 weeks
  Survey assessing daily function; scores range from 0 to 53 for the ADL section and 0 to 16 for the instrumental ADL section, with lower scores demonstrating more functional impairment.
Alzheimer's Disease Cooperative Scale - Clinical Global Impression of Change (ADCS-MCI-CGIC) score | Change from baseline at 12 and 24 weeks
  Clinical assessment of global function. The Clinician's Global Impression of Change Scale (ADCS-MCI-CGIC) is rated on a 7-point scale with the change scale using a range of responses from 1 (very much improved) through 7 (very much worse).
Neuropsychiatric Inventory (NPI) sub score | Change from baseline at 12 and 24 weeks
  Informant interview assessment of patient's neuropsychiatric symptom severity. The score for each domain is defined as frequency times severity and total NPI score is defined as the sum of the individual category scores. Higher scores on NPI indicate a more frequent and/or severe presence of neuropsychiatric behavioral changes. The following domains will be included in the subscore: Depression/Dysphoria, Anxiety, Apathy/Indifference, Irritability/Lability, Agitation/Aggression, and Disinhibition.

OTHER OUTCOMES:
Physical Activity Scale for the Elderly (PASE) | Change from baseline at 12 and 24 weeks
  The PASE is a short survey designed to assess physical activity specifically in elderly.
Geriatric Depression Scale (GDS) | Change from baseline at 12 and 24 weeks
  The GDS is a self-report measure of depression in older adults. Users respond to 30 questions in a "Yes/No" format. In scoring the GDS, each item is scored 0 or 1 depending upon whether the item is worded positively or negatively. The total score on the scale ranges from 0 to 30.
Brief Smell Identification Test (BSIT) score | Change from baseline at 12 and 24 weeks
  Olfaction assessment. The total olfaction score is defined as the number of odorants correctly identified out of the 12 tested, with higher scores denoting better performance. Identification of fewer than nine odorants is considered abnormal olfactory function.
Neuropsychiatric Inventory (NPI) total score | Change from baseline at 12 and 24 weeks
  Informant interview assessment of patient's neuropsychiatric symptom severity. The score for each domain is defined as frequency times severity and total NPI score is defined as the sum of the individual category scores. Higher scores on NPI indicate a more frequent and/or severe presence of neuropsychiatric behavioral changes.
Neuropsychological Test Battery (NTB) standardized composite score at 12 weeks | 12 weeks
  Standardized composite score generated from a battery of 4 cognitive tests, including: 1) COWAT - Category Fluency assessment of semantic fluency; 2) WAIS-IV Coding (Digit Symbol Substitution Test; DSST) assesment of attention speed of processing, mental flexibility and executive function; 3) Free and Cued Selective Reminding Test Immediate Recall (FCSRT-IR) assessment of episodic visual memory; 4) Wechsler Logical Memory II (Delayed Recall) assessment of narrative memory.
Clinical Dementia Rating Scale - Sum of Boxes (CDR-SB) score at 12 weeks | 12 weeks
  Composite measure of cognition and global function. The scores in each domain range from 0-3, referring to impairment with 0 being none, 0.5 being questionable, 1 being mild, 2 being moderate, and 3 being severe.
Responder analyses of Modified Mini-Mental State Examination (mMMSE) | Change from baseline at 12 and 24 weeks
  Cognitive test; the mMMSE is scored as the number of correctly completed items, with lower scores indicative of poorer performance and greater cognitive impairment. The score ranges from 0 to 100, with 100 being perfect performance. Positive responders are subjects who achieve at least a 3-point improvement on mMMSE
Neuropsychological Test Battery cognitive domain analyses | Change from baseline at 12 and 24 weeks, or change from baseline at 24 weeks, as appropriate
  Analysis of individual cognitive tests comprising the Neuropsychological Test Battery (NTB)
Insulin resistance markers | Change from baseline at 12 and 24 weeks
  HbA1c and Homeostatic Model Assessment of Insulin Resistance (HOMA-IR): fasting glucose and insulin

CONTACTS AND LOCATIONS:
Overall Officials: Douglas W Scharre, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No